CLINICAL TRIAL: NCT02998866
Title: Cryoballoon Pulmonary Vein Isolation and Associated Esophageal Effects
Brief Title: Cryoballoon Pulmonary Vein Isolation Including Associated Esophageal Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI1002BD
Record Dates: First submitted 2016-11-18; First posted 2016-12-21 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2016-12

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Cryoballoon Pulmonary Vein Isolation; Esophageal Effects
MeSH Terms: conditions — Atrial Fibrillation

ARMS (1):
- Multi-center, prospective outcomes registry (Other): The study is a multi-center, prospective outcomes registry
  Interventions: Procedure: Esophageal Temperature-Guided Ablation

INTERVENTIONS:
Procedure: Esophageal Temperature-Guided Ablation — Esophageal temperature-guided ablation (if esophageal temperatures drop too low during cryoablation, the physician will stop the ablation) in order to increase the safety profile of cryoballoon pulmonary vein (a vein carrying blood from the participants lungs to the left side of the participants heart known as the left atrium) isolation (PVI [means a balloon shaped catheter will be placed at the opening of each pulmonary vein and tissue will be cooled in order to create an ablation line (line of scar tissue) between the left side of the participants heart and each pulmonary vein. This is done to prevent the triggers that typically cause intermittent atrial fibrillation (known as Paroxsymal Atrial Fibrillation) by providing one center's experience.

SUMMARY:
To determine the correlation between rate of temperature decline and nadir cryoballoon temperatures rate of temperature decline and nadir esophageal temperatures during pulmonary vein isolation.

DETAILED DESCRIPTION:
When treating atrial fibrillation and targeting various areas in the left atrium, electrophysiologists have the choice to perform ablation with RF energy or cryoenergy. Esophageal ulceration and in more rare cases, esophageal fistulae, are known complications of this ablation procedure. Though rare (0.1-0.25% fistula rate and 15-20% esophageal ulceration rate according to the most recent Heart Rhythm Society EHRA ECA consensus statement)1, the investigators would very much like to understand how to completely prevent these occurrences. Cryoenergy has more recently been introduced as an energy source used in the PVI procedure; therefore, for this energy source, rates of esophageal ulceration are not yet well-defined. Nine esophageal fistulae have occurred in the first approximately 130,000 cryoballoon procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent, symptomatic, drug-refractory, paroxysmal atrial fibrillation with planned cryoballoon pulmonary vein isolation
2. Age >18 years
3. Planned AF cryoablation procedure

Exclusion Criteria:

1. LA diameter >55mm
2. Severe LVH (LV wall ≥ 15mm)
3. LA thrombus
4. Decompensated heart failure
5. Plans for left atrial ablation lesions beyond isolation of the pulmonary veins
6. History of previous pulmonary vein isolation
7. Inability to place esophageal temperature probe or TEE probe
8. Previously documented phrenic nerve injury
9. Known esophageal pathology (complete GI history worksheet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11; Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Temperature Decline | 90 days or when complications resolve
  I. To determine the correlation between rate of temperature decline and nadir cryoballoon temperatures rate of temperature decline and nadir esophageal temperatures during pulmonary vein isolation procedure.
Measurements of esophagus to each pulmonary vein | 90 days or when complications resolve
  II. To accurately measure the distance between the esophagus and the ostium of each pulmonary vein intra-operatively.
Create Recommendations for esophageal temperature-guided ablation | 90 days or when complications resolve
  To attempt to create recommendations for esophageal temperature-guided ablation in order to increase the safety profile of cryoballoon pulmonary vein isolation (PVI) by providing one center's experience. By trending cryoballoon ablation temperatures and subsequent esophageal temperatures, data trends may emerge and be predictive for esophageal ulceration formation. These trends may include:
  * Distance between esophagus and pulmonary vein in patients who developed post-ablation esophageal ulcerations
  * Intra-procedure esophageal temperatures in patients who developed post-ablation esophageal ulcerations
  * Intra-procedure cryoballoon temperatures in patients who developed post-ablation esophageal ulcerations
Assessment of additional Adverse Events | 90 days or when complications resolve
  To associate the development of symptoms (including dysphagia, chest pain, fever, "heartburn," or odynophagia) with the presence of ulcerations.

SECONDARY OUTCOMES:
Data collection on Phrenic Injury | 90 days or when complications resolve
  Assess participants with abnormal imaging and/or adverse events that are related to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Deville, MD, Principal Investigator — The Heart Hospital Baylor of Plano